CLINICAL TRIAL: NCT03394144
Title: A Phase I, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AZD9150 Monotherapy and AZD9150 in Combination With Durvalumab in Japanese Patients With Advanced Solid Malignancies
Brief Title: Study of AZD9150 and MEDI4736 (Durvalumab) in Japanese Adult Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5660C00017
Record Dates: First submitted 2017-11-10; First posted 2018-01-09 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — danvatirsen; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C1:AZD9150, C2:AZD9150+Durvalumab (Experimental): After confirmed safety with Cohort 1, Cohort 2 will open
  Interventions: Drug: AZD9150, Durvalumab

INTERVENTIONS:
Drug: AZD9150, Durvalumab — After confirmed safety with Cohort 1, Cohort 2 will open. Patients allocated in each cohort will be evaluated for DLT

SUMMARY:
This is a phase I, open-label study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of AZD9150 monotherapy and AZD9150 in combination with durvalumab in Japanese patients with advanced solid malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients must be at least 20 years of age.
* Has an Eastern Cooperative Oncology Group (ECOG) PS score of 0 or 1.
* Has measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) with a minimum size of 10 mm by computerised tomography (CT) scan, except lymph nodes which must have minimum short axis size of 15 mm (CT scan slice thickness no greater than 5 mm in both cases).
* Adequate organ and marrow function
* Female subjects of childbearing potential and male subjects with partners of childbearing potential should ensure use of a highly effective method of birth control as defined in study protocol

Key Exclusion Criteria:

* Spinal cord compression unless asymptomatic and not requiring steroids for at least 4 weeks before the start of study treatment.
* Patients must have completed any previous cancer-related treatments before enrolment.
* Has active or prior autoimmune disease within the past 2 years
* Has active or prior inflammatory bowel disease or primary immunodeficiency
* Undergone an organ transplant that requires use of immunosuppressive treatment
* Abnormalities in rhythm, conduction or morphology of resting 12-lead ECG
* Prior exposure to AZD9150 or any other anti PD (L)1 antibody.

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in terms of adverse events | From obtaining the first informed consent until 28 days after the last dose (AZD9150). In patients with Durvalumab until 90 days after the last dose (Durvalumab). Expected to be for up to 12 months.
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From obtaining the first informed consent until 28 days after the last dose (AZD9150). In patients with Durvalumab for 90 days for the last dose (Durvalumab). Expected to be for up to 12 months.
  Pharmacokinetics (PK) parameters will be derived using standard non-compartmental methods.
Overall response rate | Assessed at every even numbered cycle with RECIST until disease progression. Expected to be for up to 12 months.
  Defined as the proportion of subjects who achieve a response.
Duration of Response | Assessed at every even numbered cycle with RECIST until disease progression. Expected to be for up to 12 months.
  Defined as the interval from the first documentation of response to the earlier of the first documentation of definitive disease progression or death from any cause.
Area under the plasma concentration-time curve (AUC) | From obtaining the first informed consent until 28 days after the last dose (AZD9150). In patients with Durvalumab for 90 days for the last dose (Durvalumab). Expected to be for up to 12 months.
  PK parameters will be derived using standard non-compartmental methods.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research Site, Kashiwa
  - Research Site, Matsuyama

REFERENCES:
- [Derived] Nishina T, Fujita T, Yoshizuka N, Sugibayashi K, Murayama K, Kuboki Y. Safety, tolerability, pharmacokinetics and preliminary antitumour activity of an antisense oligonucleotide targeting STAT3 (danvatirsen) as monotherapy and in combination with durvalumab in Japanese patients with advanced solid malignancies: a phase 1 study. BMJ Open. 2022 Oct 21;12(10):e055718. doi: 10.1136/bmjopen-2021-055718. PMID 36270753